CLINICAL TRIAL: NCT00000542
Title: Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 85; P20RR011104 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2009-02

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Diabetes Mellitus; Heart Diseases; Hypercholesterolemia; Hypertension; Myocardial Infarction; Myocardial Ischemia; Heart Failure
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Diabetes Mellitus; Heart Diseases; Hypercholesterolemia; Hypertension; Myocardial Infarction; Myocardial Ischemia; Heart Failure | interventions — Angiotensin-Converting Enzyme Inhibitors; Amlodipine; Lisinopril; Doxazosin; Chlorthalidone; Pravastatin; Diet, Fat-Restricted

INTERVENTIONS:
Drug: Inhibitors, ACE
Drug: amlodipine
Drug: lisinopril
Drug: doxazosin
Drug: chlorthalidone
Drug: pravastatin
Behavioral: diet, fat-restricted

SUMMARY:
To determine if the combined incidence of nonfatal myocardial infarction and coronary heart disease death differs between diuretic-based and each of three alternative antihypertensive pharmacological treatments. Also, to determine, in a subset of this population, if lowering serum cholesterol with a HMG CoA reductase inhibitor in older adults reduces all-cause mortality compared to a control group receiving usual care. Conducted in conjunction with the Department of Veterans' Affairs.

DETAILED DESCRIPTION:
BACKGROUND:

An estimated 58 million people in the United States have elevated blood pressure (systolic blood pressure (SBP) of 140 mmHg or greater and/or diastolic blood pressure (DBP) of 90 mmHg or greater on initial examination) or are taking antihypertensive medication. Perhaps one-half to two-thirds of these have sustained hypertension.

Despite the known etiologic relationship of hypertension to coronary heart disease, large-scale randomized clinical trials in mild to moderate hypertension have failed to demonstrate conclusively that antihypertensive drug treatment, largely based on thiazide-like diuretics, reduces the occurrence of coronary heart disease death or non-fatal myocardial infarction. The pooled results of nine such trials, using primarily thiazide-like diuretics and involving over 43,000 subjects, suggest a 9 percent benefit, with 95 percent confidence limits consistent with a 19 percent benefit or 1 percent adverse outcome. This observed treatment effect compares with a maximum predicted effect on coronary heart disease of approximately 23 percent for an equivalent blood pressure difference, as derived from epidemiologic data. In contrast, the observed beneficial effect on stroke in these trials, 36 percent, is almost exactly that which would be predicted from epidemiologic data. A more recent overview of 14 trials in participants with all levels of hypertension estimated a somewhat larger benefit of 14 percent. While this may be an over-estimate of benefit, these overviews do not include the strongly positive results of the Systolic Hypertension in the Elderly Program (SHEP), in which diuretic-based treatment reduced stroke incidence by 36 percent and major coronary heart disease events by 27 percent.

In the early 1980s, two new classes of antihypertensive agents, the calcium antagonists and ACE inhibitors, were developed and licensed for use in chronic antihypertensive therapy. These agents cost more than older agents such as diuretics and beta-blockers, and evidence was limited that might justify their use despite the increased cost. The 1988 Joint National Committee on Detection, Evaluation, and Treatment of High Blood Pressure recommended beta-blockers, calcium antagonists, ACE-inhibitors, and diuretics as equally acceptable first-line therapy. All four classes of drugs have been found to control diastolic blood pressure as single agents in 50 percent or more of patients with mild hypertension.

Of these drug classes, only beta-blockers have been compared directly to diuretics in large-scale, long-term clinical trials in hypertension. Three such trials completed in Europe in 1985-1986 showed approximate equivalence of effects on morbidity and mortality in diuretic- and beta-blocker-based regimens. Pooled analysis of these trials yields a 6 percent lower coronary heart disease mortality from beta-blockers. These data are in contrast to the recent Medical Research Council (MRC) Trial in the Elderly, in which patients treated with a thiazide diuretic had significantly lower rates of coronary heart disease compared to beta-blocker treatment or placebo, both by about 45 percent.

Circulating levels of cholesterol, specifically cholesterol associated with the low-density lipoprotein (LDL) fraction, have been established as a major etiologic factor in coronary heart disease in observational epidemiologic studies, in metabolic, pathologic, and genetic studies in humans and selected animal models, and in randomized clinical trials. The clinical trials that have demonstrated a reduction in coronary heart disease incidence from lowering LDL-cholesterol levels have been conducted primarily in middle-aged men with hypercholesterolemia or established coronary heart disease. Experimental evidence for the efficacy of cholesterol lowering in older men is confined to the analysis of small subgroups of clinical trials and is lacking for women of any age. The paucity of clinical trial data led the National Cholesterol Education Program's Expert Panel on Detection, Evaluation, and Treatment of High Blood Cholesterol in Adults in their 1987 Guidelines to allow for considerable physician judgement regarding the elderly.

DESIGN NARRATIVE:

Patients were recruited through office-based practices and hypertension clinics which were reimbursed by the Clinical Trials Center on a per-patient basis. Six hundred patients were entered into the vanguard or feasibility phase and a total of 42,448 were entered into the full-scale trial. The primary hypothesis of the antihypertensive trial was that the combined incidence of fatal coronary heart disease and nonfatal myocardial infarction would be lower in hypertensive patients randomized to amlodipine (a calcium antagonist), lisinopril (an angiotensin-converting enzyme (ACE) inhibitor), or doxazosin (an alpha adrenergic blocker) as compared to those randomized to chlorthalidone (a thiazide-like diuretic). Secondary endpoints were total cardiovascular mortality, major morbidity, all-cause mortality, and health-related quality of life.

The primary hypothesis of the cholesterol-lowering trial was that mortality from all causes would be lower in the subset of hypertensive patients with LDL cholesterol levels between 120 and 189 mg/dl (between 100 and 159 mg/dl for those with known coronary heart disease) who were randomized to receive pravastatin (a HMG CoA reductase inhibitor) plus the National Cholesterol Education Program Step I cholesterol-lowering diet than those randomized to receive usual care plus diet. Secondary endpoints were the combined incidence of nonfatal myocardial infarction and coronary heart disease death, major non-cardiovascular heart disease morbidity and mortality, and health-related quality of life.

Recruitment for the feasibility phase began in February 1994. The clinical phase of the feasibility study ended in September 1994. Recruitment for the full-scale trial began in October 1994 and ended in January, 1998. The mean follow-up was 4.9 years. There were over 600 clinics in 47 states, Puerto Rico, Virgin Islands and Canada.

ELIGIBILITY:
Men and women hypertensive patients, ages 55 and above. A total of 36 percent were diabetics.

Ages: 55 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1993-08; Primary Completion 2002-03 (Actual); Study Completion 2002-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry Davis — University of Texas

REFERENCES:
- [Background] Whelton PK, Williamson JD, Louis GT, Davis BR, Cutler JA. Experimental approaches to determining the choice of first-step therapy for patients with hypertension. The ALLHAT Research Group Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Clin Exp Hypertens. 1996 Apr-May;18(3-4):569-79. doi: 10.3109/10641969609088986. PMID 8743044
- [Background] Elliott WJ. ALLHAT: the largest and most important clinical trial in hypertension ever done in the USA. Antihypertensive and Lipid Lowering Treatment to Prevent Heart Attack Trial. Am J Hypertens. 1996 Apr;9(4 Pt 1):409-11. No abstract available. PMID 8722446
- [Background] Saunders E. Recruitment of African-American patients for clinical trials--the Allhat challenges. Antihypertensive and Lipid-lowering Trial to Prevent Heart Attack. J Natl Med Assoc. 1995 Aug;87(8 Suppl):627-9. No abstract available. PMID 7674359
- [Background] Manolio TA, Cutler JA, Furberg CD, Psaty BM, Whelton PK, Applegate WB. Trends in pharmacologic management of hypertension in the United States. Arch Intern Med. 1995 Apr 24;155(8):829-37. PMID 7717791
- [Background] Davis BR, Cutler JA, Gordon DJ, Furberg CD, Wright JT Jr, Cushman WC, Grimm RH, LaRosa J, Whelton PK, Perry HM, Alderman MH, Ford CE, Oparil S, Francis C, Proschan M, Pressel S, Black HR, Hawkins CM. Rationale and design for the Antihypertensive and Lipid Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). ALLHAT Research Group. Am J Hypertens. 1996 Apr;9(4 Pt 1):342-60. doi: 10.1016/0895-7061(96)00037-4. PMID 8722437
- [Background] Conlin PR, Williams GH. Use of calcium channel blockers in hypertension. Adv Intern Med. 1998;43:533-62. PMID 9506192
- [Background] Anderson RJ, Alonso K. The ALLHAT challenges. J Natl Med Assoc. 1996 Jun;88(6):335, 368. No abstract available. PMID 8691491
- [Background] Messerli FH. What, if anything, is controversial about calcium antagonists? Am J Hypertens. 1996 Dec;9(12 Pt 2):177S-181S. doi: 10.1016/s0895-7061(96)00387-1. PMID 8968430
- [Background] Proschan M, Davis B, Cutler J, Ford C, Furberg C, Grimm R, Oparil S. ALLHAT and calcium channel blockers. ALLHAT Research Group. Am J Hypertens. 1997 Jan;10(1):142-3. No abstract available. PMID 9008261
- [Background] Cutler JA. Calcium-channel blockers for hypertension--uncertainty continues. N Engl J Med. 1998 Mar 5;338(10):679-81. doi: 10.1056/NEJM199803053381009. No abstract available. PMID 9486999
- [Background] SoRelle R. National Heart, Lung, and Blood Institute halts part of antihypertensive and lipid-lowering treatment to prevent heart attack trial (ALLHAT). Circulation. 2000 Mar 28;101(12):E9025. doi: 10.1161/01.cir.101.12.e9025. No abstract available. PMID 10736305
- [Background] Messerli FH. Implications of discontinuation of doxazosin arm of ALLHAT. Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Lancet. 2000 Mar 11;355(9207):863-4. doi: 10.1016/s0140-6736(00)00092-1. No abstract available. PMID 10752699
- [Background] Major cardiovascular events in hypertensive patients randomized to doxazosin vs chlorthalidone: the antihypertensive and lipid-lowering treatment to prevent heart attack trial (ALLHAT). ALLHAT Collaborative Research Group. JAMA. 2000 Apr 19;283(15):1967-75. PMID 10789664
- [Background] Lasagna L. Diuretics vs alpha-blockers for treatment of hypertension: lessons from ALLHAT. Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. JAMA. 2000 Apr 19;283(15):2013-4. doi: 10.1001/jama.283.15.2013. No abstract available. PMID 10789671
- [Background] Pressel SL, Davis BR, Wright JT, Geraci TS, Kingry C, Ford CE, Piller LB, Bettencourt J, Kimmel B, Lusk C, Parks H, Simpson LM, Nwachuku C, Furberg CD; ALLHAT Collaborative Research Group. Operational aspects of terminating the doxazosin arm of The Antihypertensive and Lipid Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Control Clin Trials. 2001 Feb;22(1):29-41. doi: 10.1016/s0197-2456(00)00109-4. PMID 11165421
- [Background] Grimm RH Jr, Margolis KL, Papademetriou V V, Cushman WC, Ford CE, Bettencourt J, Alderman MH, Basile JN, Black HR, DeQuattro V V, Eckfeldt J, Hawkins CM, Perry HM Jr, Proschan M. Baseline Characteristics of Participants in the Antihypertensive and Lipid Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Hypertension. 2001 Jan;37(1):19-27. doi: 10.1161/01.hyp.37.1.19. PMID 11208751
- [Background] Barzilay JI, Jones CL, Davis BR, Basile JN, Goff DC Jr, Ciocon JO, Sweeney ME, Randall OS; Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). ALLHAT Collaborative Research Group. Baseline characteristics of the diabetic participants in the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Diabetes Care. 2001 Apr;24(4):654-8. doi: 10.2337/diacare.24.4.654. PMID 11315826
- [Background] Wright JT Jr, Cushman WC, Davis BR, Barzilay J, Colon P, Egan D, Lucente T, Nwachuku C, Pressel S, Leenen FH, Frolkis J, Letterer R, Walsh S, Tobin JN, Deger GE; ALLHAT Research Group. The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT): clinical center recruitment experience. Control Clin Trials. 2001 Dec;22(6):659-73. doi: 10.1016/s0197-2456(01)00176-3. PMID 11738122
- [Background] Pressel S, Davis BR, Louis GT, Whelton P, Adrogue H, Egan D, Farber M, Payne G, Probstfield J, Ward H; ALLHAT Research Group. Participant recruitment in the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Control Clin Trials. 2001 Dec;22(6):674-86. doi: 10.1016/s0197-2456(01)00177-5. PMID 11738123
- [Background] Cushman WC, Ford CE, Cutler JA, Margolis KL, Davis BR, Grimm RH, Black HR, Hamilton BP, Holland J, Nwachuku C, Papademetriou V, Probstfield J, Wright JT Jr, Alderman MH, Weiss RJ, Piller L, Bettencourt J, Walsh SM; ALLHAT Collaborative Research Group. Success and predictors of blood pressure control in diverse North American settings: the antihypertensive and lipid-lowering treatment to prevent heart attack trial (ALLHAT). J Clin Hypertens (Greenwich). 2002 Nov-Dec;4(6):393-404. doi: 10.1111/j.1524-6175.2002.02045.x. PMID 12461301
- [Background] Piller LB, Davis BR, Cutler JA, Cushman WC, Wright JT Jr, Williamson JD, Leenen FH, Einhorn PT, Randall OS, Golden JS, Haywood LJ; The ALLHAT Collaborative Research Group. Validation of Heart Failure Events in the Antihypertensive and Lipid Lowering Treatment to Prevent Heart Attack Trial (ALLHAT) Participants Assigned to Doxazosin and Chlorthalidone. Curr Control Trials Cardiovasc Med. 2002 Nov 14;3(1):10. doi: 10.1186/1468-6708-3-10. PMID 12459039
- [Background] Pasternak RC. The ALLHAT lipid lowering trial--less is less. JAMA. 2002 Dec 18;288(23):3042-4. doi: 10.1001/jama.288.23.3042. No abstract available. PMID 12479771
- [Background] Appel LJ. The verdict from ALLHAT--thiazide diuretics are the preferred initial therapy for hypertension. JAMA. 2002 Dec 18;288(23):3039-42. doi: 10.1001/jama.288.23.3039. No abstract available. PMID 12479770
- [Background] ALLHAT Officers and Coordinators for the ALLHAT Collaborative Research Group. The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Major outcomes in moderately hypercholesterolemic, hypertensive patients randomized to pravastatin vs usual care: The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT-LLT). JAMA. 2002 Dec 18;288(23):2998-3007. doi: 10.1001/jama.288.23.2998. PMID 12479764
- [Background] ALLHAT Officers and Coordinators for the ALLHAT Collaborative Research Group. The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Major outcomes in high-risk hypertensive patients randomized to angiotensin-converting enzyme inhibitor or calcium channel blocker vs diuretic: The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). JAMA. 2002 Dec 18;288(23):2981-97. doi: 10.1001/jama.288.23.2981. PMID 12479763
- [Background] Flack JM, Nasser SA; Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT. The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Major outomes in high-risk hypertensive patients randomized to angiotensin-converting enzyme inhibitor or calcium channel blocker vs diuretic. Curr Hypertens Rep. 2003 Jun;5(3):189-91. doi: 10.1007/s11906-003-0019-8. No abstract available. PMID 12724049
- [Background] Papademetriou V, Piller LB, Ford CE, Gordon D, Hartney TJ, Geraci TS, Reisin E, Sumner BM, Wong ND, Nwachuku C, Narayan P, Haywood J, Habib G; ALLHAT Collaborative Research Group. Characteristics and lipid distribution of a large, high-risk, hypertensive population: the lipid-lowering component of the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). J Clin Hypertens (Greenwich). 2003 Nov-Dec;5(6):377-84. doi: 10.1111/j.1524-6175.2003.03163.x. PMID 14688492
- [Background] Rahman M, Brown CD, Coresh J, Davis BR, Eckfeldt JH, Kopyt N, Levey AS, Nwachuku C, Pressel S, Reisin E, Walworth C; Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial Collaborative Research Group. The prevalence of reduced glomerular filtration rate in older hypertensive patients and its association with cardiovascular disease: a report from the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Arch Intern Med. 2004 May 10;164(9):969-76. doi: 10.1001/archinte.164.9.969. PMID 15136305
- [Background] Berecek KH, Farag A, Bahtiyar G, Rothman J, McFarlane SI. The Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack (ALLHAT) Trial: focus on the diabetic patient. Curr Hypertens Rep. 2004 Jun;6(3):212-4. No abstract available. PMID 15128474
- [Background] Barzilay JI, Davis BR, Bettencourt J, Margolis KL, Goff DC Jr, Black H, Habib G, Ellsworth A, Force RW, Wiegmann T, Ciocon JO, Basile JN; ALLHAT Collaborative Research Group. Cardiovascular outcomes using doxazosin vs. chlorthalidone for the treatment of hypertension in older adults with and without glucose disorders: a report from the ALLHAT study. J Clin Hypertens (Greenwich). 2004 Mar;6(3):116-25. doi: 10.1111/j.1524-6175.2004.03216.x. PMID 15010644
- [Background] Davis BR, Furberg CD, Wright JT Jr, Cutler JA, Whelton P; ALLHAT Collaborative Research Group. ALLHAT: setting the record straight. Ann Intern Med. 2004 Jul 6;141(1):39-46. doi: 10.7326/0003-4819-141-1-200407060-00013. PMID 15238369
- [Background] Geraci TS, Geraci SA. What ALLHAT tells us about treating high-risk patients with hypertension and hyperlipidemia. J Cardiovasc Nurs. 2003 Nov-Dec;18(5):389-95. doi: 10.1097/00005082-200311000-00011. PMID 14680343
- [Background] Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial Collaborative Research Group. Diuretic versus alpha-blocker as first-step antihypertensive therapy: final results from the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Hypertension. 2003 Sep;42(3):239-46. doi: 10.1161/01.HYP.0000086521.95630.5A. Epub 2003 Aug 18. PMID 12925554
- [Background] Davis BR, Cutler JA, Furberg CD, Wright JT, Farber MA, Felicetta JV, Stokes JD; ALLHAT Collaborative Research Group. Relationship of antihypertensive treatment regimens and change in blood pressure to risk for heart failure in hypertensive patients randomly assigned to doxazosin or chlorthalidone: further analyses from the Antihypertensive and Lipid-Lowering treatment to prevent Heart Attack Trial. Ann Intern Med. 2002 Sep 3;137(5 Part 1):313-20. doi: 10.7326/0003-4819-137-5_part_1-200209030-00006. PMID 12204014
- [Background] Wright JT Jr, Dunn JK, Cutler JA, Davis BR, Cushman WC, Ford CE, Haywood LJ, Leenen FH, Margolis KL, Papademetriou V, Probstfield JL, Whelton PK, Habib GB; ALLHAT Collaborative Research Group. Outcomes in hypertensive black and nonblack patients treated with chlorthalidone, amlodipine, and lisinopril. JAMA. 2005 Apr 6;293(13):1595-608. doi: 10.1001/jama.293.13.1595. PMID 15811979
- [Background] Rahman M, Pressel S, Davis BR, Nwachuku C, Wright JT Jr, Whelton PK, Barzilay J, Batuman V, Eckfeldt JH, Farber M, Henriquez M, Kopyt N, Louis GT, Saklayen M, Stanford C, Walworth C, Ward H, Wiegmann T. Renal outcomes in high-risk hypertensive patients treated with an angiotensin-converting enzyme inhibitor or a calcium channel blocker vs a diuretic: a report from the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Arch Intern Med. 2005 Apr 25;165(8):936-46. doi: 10.1001/archinte.165.8.936. PMID 15851647
- [Background] Whelton PK, Barzilay J, Cushman WC, Davis BR, Iiamathi E, Kostis JB, Leenen FH, Louis GT, Margolis KL, Mathis DE, Moloo J, Nwachuku C, Panebianco D, Parish DC, Pressel S, Simmons DL, Thadani U; ALLHAT Collaborative Research Group. Clinical outcomes in antihypertensive treatment of type 2 diabetes, impaired fasting glucose concentration, and normoglycemia: Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Arch Intern Med. 2005 Jun 27;165(12):1401-9. doi: 10.1001/archinte.165.12.1401. PMID 15983290
- [Background] Rahman M, Pressel S, Davis BR, Nwachuku C, Wright JT Jr, Whelton PK, Barzilay J, Batuman V, Eckfeldt JH, Farber MA, Franklin S, Henriquez M, Kopyt N, Louis GT, Saklayen M, Stanford C, Walworth C, Ward H, Wiegmann T; ALLHAT Collaborative Research Group. Cardiovascular outcomes in high-risk hypertensive patients stratified by baseline glomerular filtration rate. Ann Intern Med. 2006 Feb 7;144(3):172-80. doi: 10.7326/0003-4819-144-3-200602070-00005. PMID 16461961
- [Derived] Yamal JM, Martinez J, Osani MC, Du XL, Simpson LM, Davis BR. Mortality and Morbidity Among Individuals With Hypertension Receiving a Diuretic, ACE Inhibitor, or Calcium Channel Blocker: A Secondary Analysis of a Randomized Clinical Trial. JAMA Netw Open. 2023 Dec 1;6(12):e2344998. doi: 10.1001/jamanetworkopen.2023.44998. PMID 38048133
- [Derived] Khayyat-Kholghi M, Oparil S, Davis BR, Tereshchenko LG. Worsening Kidney Function Is the Major Mechanism of Heart Failure in Hypertension: The ALLHAT Study. JACC Heart Fail. 2021 Feb;9(2):100-111. doi: 10.1016/j.jchf.2020.09.006. Epub 2020 Nov 11. PMID 33189627
- [Derived] Juraschek SP, Simpson LM, Davis BR, Shmerling RH, Beach JL, Ishak A, Mukamal KJ. The effects of antihypertensive class on gout in older adults: secondary analysis of the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. J Hypertens. 2020 May;38(5):954-960. doi: 10.1097/HJH.0000000000002359. PMID 31977576
- [Derived] Lachin JM, Bebu I. Closed testing of each group versus the others combined in a multiple group analysis. Clin Trials. 2020 Feb;17(1):77-86. doi: 10.1177/1740774519879932. Epub 2019 Oct 24. PMID 31647326
- [Derived] Juraschek SP, Simpson LM, Davis BR, Beach JL, Ishak A, Mukamal KJ. Effects of Antihypertensive Class on Falls, Syncope, and Orthostatic Hypotension in Older Adults: The ALLHAT Trial. Hypertension. 2019 Oct;74(4):1033-1040. doi: 10.1161/HYPERTENSIONAHA.119.13445. Epub 2019 Sep 3. PMID 31476905
- [Derived] Shahu A, Herrin J, Dhruva SS, Desai NR, Davis BR, Krumholz HM, Spatz ES. Disparities in Socioeconomic Context and Association With Blood Pressure Control and Cardiovascular Outcomes in ALLHAT. J Am Heart Assoc. 2019 Aug 6;8(15):e012277. doi: 10.1161/JAHA.119.012277. Epub 2019 Jul 31. PMID 31362591
- [Derived] Johnson K, Oparil S, Davis BR, Tereshchenko LG. Prevention of Heart Failure in Hypertension-Disentangling the Role of Evolving Left Ventricular Hypertrophy and Blood Pressure Lowering: The ALLHAT Study. J Am Heart Assoc. 2019 Apr 16;8(8):e011961. doi: 10.1161/JAHA.119.011961. PMID 30943832
- [Derived] Lai D, Zhang Q, Yamal JM, Einhorn PT, Davis BR; ALLHAT Collaborative Research Group. Conditional moving linear regression: modeling the recruitment process for ALLHAT. Commun Stat Theory Methods. 2017;46(18):8943-8951. doi: 10.1080/03610926.2016.1197251. Epub 2017 May 19. PMID 30906106
- [Derived] Barzilay JI, Lai D, Davis BR, Pressel S, Previn HE, Arnett DK. The Interaction of a Diabetes Gene Risk Score With 3 Different Antihypertensive Medications for Incident Glucose-level Elevation. Am J Hypertens. 2019 Mar 16;32(4):343-349. doi: 10.1093/ajh/hpy199. PMID 30590387
- [Derived] Barzilay JI, Davis BR, Ghosh A, Pressel SL, Rahman M, Einhorn PT, Cushman WC, Whelton PK, Wright JT Jr; ALLHAT Collaborative Research Group. Rapid eGFR change as a determinant of cardiovascular and renal disease outcomes and of mortality in hypertensive adults with and without type 2 diabetes. J Diabetes Complications. 2018 Sep;32(9):830-832. doi: 10.1016/j.jdiacomp.2018.07.003. Epub 2018 Jul 11. PMID 30030011
- [Derived] Itoga NK, Tawfik DS, Lee CK, Maruyama S, Leeper NJ, Chang TI. Association of Blood Pressure Measurements With Peripheral Artery Disease Events. Circulation. 2018 Oct 23;138(17):1805-1814. doi: 10.1161/CIRCULATIONAHA.118.033348. PMID 29930023
- [Derived] Dewland TA, Soliman EZ, Yamal JM, Davis BR, Alonso A, Albert CM, Simpson LM, Haywood LJ, Marcus GM. Pharmacologic Prevention of Incident Atrial Fibrillation: Long-Term Results From the ALLHAT (Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial). Circ Arrhythm Electrophysiol. 2017 Dec;10(12):e005463. doi: 10.1161/CIRCEP.117.005463. PMID 29212812
- [Derived] Shams T, Auchus AP, Oparil S, Wright CB, Wright J, Furlan AJ, Sila CA, Davis BR, Pressel S, Yamal JM, Einhorn PT, Lerner AJ; ALLHAT Collaborative Research Group. Baseline Quality of Life and Risk of Stroke in the ALLHAT Study (Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial). Stroke. 2017 Nov;48(11):3078-3085. doi: 10.1161/STROKEAHA.117.016062. Epub 2017 Sep 27. PMID 28954920
- [Derived] Han BH, Sutin D, Williamson JD, Davis BR, Piller LB, Pervin H, Pressel SL, Blaum CS; ALLHAT Collaborative Research Group. Effect of Statin Treatment vs Usual Care on Primary Cardiovascular Prevention Among Older Adults: The ALLHAT-LLT Randomized Clinical Trial. JAMA Intern Med. 2017 Jul 1;177(7):955-965. doi: 10.1001/jamainternmed.2017.1442. PMID 28531241
- [Derived] Bang CN, Soliman EZ, Simpson LM, Davis BR, Devereux RB, Okin PM; ALLHAT Collaborative Research Group. Electrocardiographic Left Ventricular Hypertrophy Predicts Cardiovascular Morbidity and Mortality in Hypertensive Patients: The ALLHAT Study. Am J Hypertens. 2017 Sep 1;30(9):914-922. doi: 10.1093/ajh/hpx067. PMID 28430947
- [Derived] Puttnam R, Davis BR, Pressel SL, Whelton PK, Cushman WC, Louis GT, Margolis KL, Oparil S, Williamson J, Ghosh A, Einhorn PT, Barzilay JI; Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT) Collaborative Research Group. Association of 3 Different Antihypertensive Medications With Hip and Pelvic Fracture Risk in Older Adults: Secondary Analysis of a Randomized Clinical Trial. JAMA Intern Med. 2017 Jan 1;177(1):67-76. doi: 10.1001/jamainternmed.2016.6821. PMID 27893045
- [Derived] Whittle J, Yamal JM, Williamson JD, Ford CE, Probstfield JL, Beard BL, Marginean H, Hamilton BP, Suhan PS, Davis BR; ALLHAT Collaborative Research Group. Clinical and demographic correlates of medication and visit adherence in a large randomized controlled trial. BMC Health Serv Res. 2016 Jul 8;16:236. doi: 10.1186/s12913-016-1471-x. PMID 27391223
- [Derived] Dewland TA, Soliman EZ, Davis BR, Magnani JW, Yamal JM, Piller LB, Haywood LJ, Alonso A, Albert CM, Marcus GM; Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT) Collaborative Research Group. Effect of the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT) on Conduction System Disease. JAMA Intern Med. 2016 Aug 1;176(8):1085-92. doi: 10.1001/jamainternmed.2016.2502. PMID 27367818
- [Derived] Kaasenbrood L, Poulter NR, Sever PS, Colhoun HM, Livingstone SJ, Boekholdt SM, Pressel SL, Davis BR, van der Graaf Y, Visseren FL; CARDS, ALLHAT, and ASCOT Investigators. Development and Validation of a Model to Predict Absolute Vascular Risk Reduction by Moderate-Intensity Statin Therapy in Individual Patients With Type 2 Diabetes Mellitus: The Anglo Scandinavian Cardiac Outcomes Trial, Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial, and Collaborative Atorvastatin Diabetes Study. Circ Cardiovasc Qual Outcomes. 2016 May;9(3):213-21. doi: 10.1161/CIRCOUTCOMES.115.001980. Epub 2016 May 11. PMID 27174798
- [Derived] Alderman MH, Davis BR, Piller LB, Ford CE, Baraniuk MS, Pressel SL, Assadi MA, Einhorn PT, Haywood LJ, Ilamathi E, Oparil S, Retta TM; ALLHAT Collaborative Research Group. Should Antihypertensive Treatment Recommendations Differ in Patients With and Without Coronary Heart Disease? (from the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial [ALLHAT]). Am J Cardiol. 2016 Jan 1;117(1):105-15. doi: 10.1016/j.amjcard.2015.10.012. Epub 2015 Oct 19. PMID 26589819
- [Derived] Yamal JM, Oparil S, Davis BR, Alderman MH, Calhoun DA, Cushman WC, Fendley HF, Franklin SS, Habib GB, Pressel SL, Probstfield JL, Sastrasinh S; ALLHAT Collaborative Research Group. Stroke outcomes among participants randomized to chlorthalidone, amlodipine or lisinopril in ALLHAT. J Am Soc Hypertens. 2014 Nov;8(11):808-19. doi: 10.1016/j.jash.2014.08.003. Epub 2014 Aug 19. PMID 25455006
- [Derived] Piller LB, Simpson LM, Baraniuk S, Habib GB, Rahman M, Basile JN, Dart RA, Ellsworth AJ, Fendley H, Probstfield JL, Whelton PK, Davis BR; ALLHAT Collaborative Research Group. Characteristics and long-term follow-up of participants with peripheral arterial disease during ALLHAT. J Gen Intern Med. 2014 Nov;29(11):1475-83. doi: 10.1007/s11606-014-2947-1. PMID 25002161
- [Derived] Reisin E, Graves JW, Yamal JM, Barzilay JI, Pressel SL, Einhorn PT, Dart RA, Retta TM, Saklayen MG, Davis BR; ALLHAT Collaborative Research Group. Blood pressure control and cardiovascular outcomes in normal-weight, overweight, and obese hypertensive patients treated with three different antihypertensives in ALLHAT. J Hypertens. 2014 Jul;32(7):1503-13; discussion 1513. doi: 10.1097/HJH.0000000000000204. PMID 24842697
- [Derived] Shah RV, Abbasi SA, Yamal JM, Davis BR, Barzilay J, Einhorn PT, Goldfine AB; ALLHAT Collaborative Research Group. Impaired fasting glucose and body mass index as determinants of mortality in ALLHAT: is the obesity paradox real? J Clin Hypertens (Greenwich). 2014 Jun;16(6):451-8. doi: 10.1111/jch.12325. Epub 2014 Apr 29. PMID 24779706
- [Derived] Phillips W, Piller LB, Williamson JD, Whittle J, Jafri SZ, Ford CE, Einhorn PT, Oparil S, Furberg CD, Grimm RH Jr, Alderman MH, Davis BR, Probstfield JL; ALLHAT Collaborative Research Group. Risk of hospitalized gastrointestinal bleeding in persons randomized to diuretic, ACE-inhibitor, or calcium-channel blocker in ALLHAT. J Clin Hypertens (Greenwich). 2013 Nov;15(11):825-32. doi: 10.1111/jch.12180. Epub 2013 Aug 7. PMID 24283598
- [Derived] Oparil S, Davis BR, Cushman WC, Ford CE, Furberg CD, Habib GB, Haywood LJ, Margolis K, Probstfield JL, Whelton PK, Wright JT Jr; ALLHAT Collaborative Research Group. Mortality and morbidity during and after Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial: results by sex. Hypertension. 2013 May;61(5):977-86. doi: 10.1161/HYPERTENSIONAHA.111.00213. Epub 2013 Mar 25. PMID 23529173
- [Derived] Drawz PE, Baraniuk S, Davis BR, Brown CD, Colon PJ Sr, Cujyet AB, Dart RA, Graumlich JF, Henriquez MA, Moloo J, Sakalayen MG, Simmons DL, Stanford C, Sweeney ME, Wong ND, Rahman M. Cardiovascular risk assessment: addition of CKD and race to the Framingham equation. Am Heart J. 2012 Dec;164(6):925-31.e2. doi: 10.1016/j.ahj.2012.09.003. Epub 2012 Oct 29. PMID 23194494
- [Derived] Rahman M, Ford CE, Cutler JA, Davis BR, Piller LB, Whelton PK, Wright JT Jr, Barzilay JI, Brown CD, Colon PJ Sr, Fine LJ, Grimm RH Jr, Gupta AK, Baimbridge C, Haywood LJ, Henriquez MA, Ilamaythi E, Oparil S, Preston R; ALLHAT Collaborative Research Group. Long-term renal and cardiovascular outcomes in Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT) participants by baseline estimated GFR. Clin J Am Soc Nephrol. 2012 Jun;7(6):989-1002. doi: 10.2215/CJN.07800811. Epub 2012 Apr 5. PMID 22490878
- [Derived] Zhang X, Lynch AI, Davis BR, Ford CE, Boerwinkle E, Eckfeldt JH, Leiendecker-Foster C, Arnett DK. Pharmacogenetic association of NOS3 variants with cardiovascular disease in patients with hypertension: the GenHAT study. PLoS One. 2012;7(3):e34217. doi: 10.1371/journal.pone.0034217. Epub 2012 Mar 28. PMID 22470539
- [Derived] Alderman MH, Piller LB, Ford CE, Probstfield JL, Oparil S, Cushman WC, Einhorn PT, Franklin SS, Papademetriou V, Ong ST, Eckfeldt JH, Furberg CD, Calhoun DA, Davis BR; Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial Collaborative Research Group. Clinical significance of incident hypokalemia and hyperkalemia in treated hypertensive patients in the antihypertensive and lipid-lowering treatment to prevent heart attack trial. Hypertension. 2012 May;59(5):926-33. doi: 10.1161/HYPERTENSIONAHA.111.180554. Epub 2012 Mar 19. PMID 22431578
- [Derived] Barzilay JI, Davis BR, Pressel SL, Cutler JA, Einhorn PT, Black HR, Cushman WC, Ford CE, Margolis KL, Moloo J, Oparil S, Piller LB, Simmons DL, Sweeney ME, Whelton PK, Wong ND, Wright JT Jr; ALLHAT Collaborative Research Group. Long-term effects of incident diabetes mellitus on cardiovascular outcomes in people treated for hypertension: the ALLHAT Diabetes Extension Study. Circ Cardiovasc Qual Outcomes. 2012 Mar 1;5(2):153-62. doi: 10.1161/CIRCOUTCOMES.111.962522. Epub 2012 Mar 6. PMID 22396585
- [Derived] Cushman WC, Davis BR, Pressel SL, Cutler JA, Einhorn PT, Ford CE, Oparil S, Probstfield JL, Whelton PK, Wright JT Jr, Alderman MH, Basile JN, Black HR, Grimm RH Jr, Hamilton BP, Haywood LJ, Ong ST, Piller LB, Simpson LM, Stanford C, Weiss RJ; ALLHAT Collaborative Research Group. Mortality and morbidity during and after the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. J Clin Hypertens (Greenwich). 2012 Jan;14(1):20-31. doi: 10.1111/j.1751-7176.2011.00568.x. Epub 2011 Dec 9. PMID 22235820
- [Derived] Piller LB, Baraniuk S, Simpson LM, Cushman WC, Massie BM, Einhorn PT, Oparil S, Ford CE, Graumlich JF, Dart RA, Parish DC, Retta TM, Cuyjet AB, Jafri SZ, Furberg CD, Saklayen MG, Thadani U, Probstfield JL, Davis BR; ALLHAT Collaborative Research Group. Long-term follow-up of participants with heart failure in the antihypertensive and lipid-lowering treatment to prevent heart attack trial (ALLHAT). Circulation. 2011 Oct 25;124(17):1811-8. doi: 10.1161/CIRCULATIONAHA.110.012575. Epub 2011 Oct 3. PMID 21969009
- [Derived] Haywood LJ, Ford CE, Crow RS, Davis BR, Massie BM, Einhorn PT, Williard A; ALLHAT Collaborative Research Group. Atrial fibrillation at baseline and during follow-up in ALLHAT (Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial). J Am Coll Cardiol. 2009 Nov 24;54(22):2023-31. doi: 10.1016/j.jacc.2009.08.020. PMID 19926008
- [Derived] Davis BR, Kostis JB, Simpson LM, Black HR, Cushman WC, Einhorn PT, Farber MA, Ford CE, Levy D, Massie BM, Nawaz S; ALLHAT Collaborative Research Group. Heart failure with preserved and reduced left ventricular ejection fraction in the antihypertensive and lipid-lowering treatment to prevent heart attack trial. Circulation. 2008 Nov 25;118(22):2259-67. doi: 10.1161/CIRCULATIONAHA.107.762229. Epub 2008 Nov 10. PMID 19001024
- [Derived] Rahman M, Baimbridge C, Davis BR, Barzilay J, Basile JN, Henriquez MA, Huml A, Kopyt N, Louis GT, Pressel SL, Rosendorff C, Sastrasinh S, Stanford C; ALLHAT Collaborative Research Group. Progression of kidney disease in moderately hypercholesterolemic, hypertensive patients randomized to pravastatin versus usual care: a report from the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Am J Kidney Dis. 2008 Sep;52(3):412-24. doi: 10.1053/j.ajkd.2008.05.027. Epub 2008 Aug 3. PMID 18676075
- [Derived] Wright JT Jr, Harris-Haywood S, Pressel S, Barzilay J, Baimbridge C, Bareis CJ, Basile JN, Black HR, Dart R, Gupta AK, Hamilton BP, Einhorn PT, Haywood LJ, Jafri SZ, Louis GT, Whelton PK, Scott CL, Simmons DL, Stanford C, Davis BR. Clinical outcomes by race in hypertensive patients with and without the metabolic syndrome: Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Arch Intern Med. 2008 Jan 28;168(2):207-17. doi: 10.1001/archinternmed.2007.66. PMID 18227370
- [Derived] Black HR, Davis B, Barzilay J, Nwachuku C, Baimbridge C, Marginean H, Wright JT Jr, Basile J, Wong ND, Whelton P, Dart RA, Thadani U; Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Metabolic and clinical outcomes in nondiabetic individuals with the metabolic syndrome assigned to chlorthalidone, amlodipine, or lisinopril as initial treatment for hypertension: a report from the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). Diabetes Care. 2008 Feb;31(2):353-60. doi: 10.2337/dc07-1452. Epub 2007 Nov 13. PMID 18000186
- [Derived] Margolis KL, Piller LB, Ford CE, Henriquez MA, Cushman WC, Einhorn PT, Colon PJ Sr, Vidt DG, Christian R, Wong ND, Wright JT Jr, Goff DC Jr; Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial Collaborative Research Group. Blood pressure control in Hispanics in the antihypertensive and lipid-lowering treatment to prevent heart attack trial. Hypertension. 2007 Nov;50(5):854-61. doi: 10.1161/HYPERTENSIONAHA.107.092650. Epub 2007 Sep 10. PMID 17846352
- [Derived] Davis BR, Piller LB, Cutler JA, Furberg C, Dunn K, Franklin S, Goff D, Leenen F, Mohiuddin S, Papademetriou V, Proschan M, Ellsworth A, Golden J, Colon P, Crow R; Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial Collaborative Research Group. Role of diuretics in the prevention of heart failure: the Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial. Circulation. 2006 May 9;113(18):2201-10. doi: 10.1161/CIRCULATIONAHA.105.544031. Epub 2006 May 1. PMID 16651474